CLINICAL TRIAL: NCT00590564
Title: SHO-SAIKO-TO for Patients With Chronic Hepatitis C Who Are Intolerant to or Have Contraindication to Interferon-Based Therapy: A Phase II Study
Brief Title: SHO-SAIKO-TO for Patients With Chronic Hepatitis C: A Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-073
Record Dates: First submitted 2007-12-21; First posted 2008-01-10 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Sho-saiko-to; SST; Interferon Therapy
MeSH Terms: conditions — Hepatitis C | interventions — shosaiko-to; Somatostatin-28

ARMS (1):
- 1 (Experimental): All patients will receive treatment with 2.5grams of SST as granules in packet form by mouth three times a day every day for 52 weeks unless occurrence of unacceptable adverse events or patient withdrawal.
  Interventions: Drug: Sho-saiko-to

INTERVENTIONS:
Drug: Sho-saiko-to — All patients will receive treatment with 2.5grams of SST as granules in packet form by mouth three times a day every day for 52 weeks unless occurrence of unacceptable adverse events or patient withdrawal. Patients will be seen for clinical follow-up at three month intervals: at 3, 6, 9, and 12 months, and assessed for compliance and asked about side effects and pulmonary symptoms. At each clinic visit, a comprehensive metabolic profile will be performed. At the 6-month clinic visit, a CBC will be performed. At the 12-month clinic visit, quantitative HCV-RNA by PCR will be obtained (Viromed Labs, Inc., 6101 Blue Circle Drive, Minneapolis, MN 5534). Within 4 weeks after the 12-month clinic visit (after 52 weeks of SST therapy), the second liver biopsy will be scheduled and performed.
  Other Names: sst

SUMMARY:
Researchers want to see whether Sho-saiko-to (SST) can help in patients with chronic hepatitis C. Chronic hepatitis C may cause swelling within the liver and this can lead to scar tissue. In some patients, severe scarring of the liver, liver failure and liver cancer can occur. Standard treatment for chronic hepatitis C is a drug called interferon with or without another drug called ribavirin. There are a number of side effects that some patients are unable to take. Other patients may have an initial response, but then the virus and the inflammation come back.

Sho-saiko-to is an herbal medicine that has been used for many years in Asia to treat liver disease. The purpose of the study is to evaluate whether Sho-saiko-to may improve liver swelling and injury caused by chronic hepatitis C.

DETAILED DESCRIPTION:
Chronic hepatitis C affects nearly three million Americans. Of these, 15% will develop liver cirrhosis and approximately 5% will progress to hepatocellular carcinoma. Treatment for chronic hepatitis C is limited to interferon-based therapy. Many patients decline or cannot tolerate interferon because of its serious side effects. Sho-saiko-to, an Asian herbal medicine consisting of seven botanicals, has demonstrated anti-fibrotic affect by inhibition of lipid peroxidation in hepatocytes and stellate cells in an animal study. It has also been demonstrated to prevent progression of cirrhosis to hepatocellular carcinoma in human trials. This study is a single arm, single center trial of Sho-saiko-to in patients with chronic active hepatitis from hepatitis C infection who cannot tolerate or who have specific contraindications to interferon therapy. Patients will receive 52 weeks therapy with Sho-saiko-to. Outcome will be assessed by comparing pre- and posttreatment liver biopsies. Patients will be said to respond if they have an improvement of two points or greater on a standard measure of liver histology. If five or more of 25 evaluable patients respond, Sho-saiko-to will be deemed worthy of further testing.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C diagnosis, with abnormal liver function tests, positive serology for Hepatitis C antibody, positive viremia as indicated by PCR techniques.
* Age 18 or over
* There must be no plans to use interferon in the following 12 months due to EITHER: a specific contraindication to interferon therapy, including but not limited to:history of depression, or other psychiatric disease, history of autoimmune disease,psoriasis, rheumatoid arthritis, history of renal dysfunction, thyroid abnormalities, seizure disorder, depressed blood cell counts, history of asthma OR patient discontinuation of interferon-based therapy prematurely due to intolerable side effects with sustained active viremia OR patient refusal to take interferon
* Patients must be able to understand and sign informed consent.
* Female participants must agree to practice approved methods of birth control (if applicable).

Exclusion Criteria:

* Coinfection with hepatitis B as defined by a positive Hepatitis B surface antigen (HBsAg) test.
* Coinfection with HIV
* Patients with alcohol intake >40g day
* Patients with recent myocardial infarction or heart failure.
* Concurrent use of Sho-saiko-to, or any of its constituent plants.
* Concurrent use of interferon containing products.
* Use of interferon-based treatment within the past 6 months.
* Women who are pregnant, nursing, or have the potential to becoming pregnant, unless utilizing birth control. A negative pregnancy test must be documented during the screening period for women of childbearing potential.
* History of malignancy, unless there is currently no evidence of disease and patient completed all surgery, radiotherapy and chemotherapy for that disease a minimum of two years previously
* Concurrent life-threatening illness, for which the prognosis is poor.
* Patients with diffusing capacity on pulmonary testing less than 50% of predicted will be excluded.
* Patients with diffusing capacity on pulmonary testing less than 70% of predicted AND total lung capacity less than 80% of predicted will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Deng, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Sho-saiko-to: All patients will receive treatment with 2.5grams of SST as granules in packet form by mouth three times a day every day for 52 weeks.
Period: Overall Study
Arm/Group | All Patients
Started | 42
Completed | 24
Not Completed | 18
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 1
Not completed — Patient Found to be Ineligible | 1
Not completed — Patient Non-compliance | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Effects of Sho-saiko-to on Hepatic Injury in Patients With Chronic Hepatitis C Who Are Intolerant or Have a Specific Contraindication to Interferon-based Therapy.
Description: Response is determined by improvement of 2 points or greater as per Knodell's histology activity index (HAI) scores in paired comparisons of pre and post liver biopsy
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 24
participants
  Responders | 5
  Non-responders | 19

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=24)
Conduction abnormality (Cardiac disorders) | 1 (1)
Cellulitis (skin) (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=24)
Abdominal pain/cramping (Gastrointestinal disorders) | 2 (2)
Bilirubin (Hepatobiliary disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Neutrophils (Blood and lymphatic system disorders) | 3 (3)
Aspartate Aminotransferase (AST) (Blood and lymphatic system disorders) | 6 (6)
Alanine Aminotransferase (ALT) (Blood and lymphatic system disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes